CLINICAL TRIAL: NCT01296594
Title: Improving Antihypertensive Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-080-3; P30DA023918 (NIH)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: High Blood Pressure; Substance Abuse
MeSH Terms: conditions — Hypertension; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care
- usual care with cell phone monitoring and CM (Experimental): In the CM condition, patients will carry a cell phone and record and send in time- and date-stamped self videos of medication ingestion.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Other: Usual Care — Usual Care
  Arms: Usual Care
Behavioral: Contingency Management — This intervention consists of congratulatory messages or reminders about adherence, and participants will earn vouchers each time medication ingestion occurs at the appropriate time, along with bonuses for sustained adherence.
  Arms: usual care with cell phone monitoring and CM

SUMMARY:
Poor adherence to antihypertensive medications is associated with morbidity, and data suggest that substance abuse may contribute to poor adherence. Contingency management (CM), an intervention highly efficacious for improving outcomes of substance abusers, shows promise in improving medication adherence in a handful of small trials. CM involves providing tangible reinforcement each time the behavior (medication ingestion) is exhibited. Thus far, studies evaluating CM for increasing medication adherence have utilized MEMS caps, but reinforcement of adherence via MEMS caps is done relatively infrequently and with delay, hindering its efficacy. A widely utilized technology that may be more appropriate for reinforcing medication adherence is cell phones, which can record the process of pill ingestion through video functions. As regular monitoring and feedback is important in the efficacy of CM, patients can be provided with daily messages regarding adherence and CM earnings. In this pilot study, we propose to randomize 40 hypertensive substance abusing patients with suboptimal adherence to antihypertensive medications to one of two 12-week treatment conditions: (1) usual care, or (2) usual care with cell phone monitoring and CM. In the CM condition, patients will carry a cell phone and record and send in time- and date-stamped self videos of medication ingestion. These patients will receive congratulatory messages or reminders about adherence, and they will earn vouchers each time medication ingestion occurs at the appropriate time, along with bonuses for sustained adherence. We hypothesize that the CM condition will improve self report and pill count measurements of medication adherence and that it will result in decreased blood pressure. Results from this study may have widespread implications for the use of cell phones as a novel technology to improve medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* have been prescribed one or more antihypertensive medications
* blood pressure of >120 mmHg systolic or >80 mmHg diastolic
* substance use problem
* willing to use a cell phone to record medication ingestion for three months
* have a valid photo ID (driver's license, passport, state ID) and are willing to sign an off-campus property transfer form and return study equipment at the end of study participation

Exclusion Criteria:

* uncontrolled psychiatric disorders
* significant cognitive impairment
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
self reports of medication adherence | month 3

SECONDARY OUTCOMES:
ambulatory (24-hour) blood pressure | month 3

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — University of Conncecticut Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States